CLINICAL TRIAL: NCT06955130
Title: Lactate and Glycerol Contribution to Gluconeogenesis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Ankit Shah, MD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2019002628
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes; Obesity; Healthy
Keywords: diabetes; glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus | interventions — Glycerol; Lactic Acid; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Glycerol (Experimental): Each subject will receive labeled 13C3-glycerol.
  Interventions: Drug: Glycerol
- Lactate (Experimental): Each subject will receive labeled 13C3-lactate.
  Interventions: Drug: Lactate
- Glucose (Experimental): Each subject will receive labeled 13C6-glucose.
  Interventions: Drug: Glucose

INTERVENTIONS:
Drug: Glycerol — Subjects will receive an infusion of glycerol and glucagon.
  Arms: Glycerol
Drug: Lactate — Subjects will receive an infusion of lactate and glucagon.
  Arms: Lactate
Drug: Glucose — Subjects will receive an infusion of glucose and glucagon.
  Arms: Glucose

SUMMARY:
A major cause of increased blood glucose levels in type 2 diabetes (T2D) is increased hepatic gluconeogenesis (GNG), as the liver converts various substrates into glucose. Two of these substrates include glycerol, a molecule from fat, and lactate, a molecule that circulates in the blood. Our previously collected data suggest that glycerol's role in this process has been underestimated, so the investigators will directly compare the carbon contribution of glycerol and lactate to new glucose production under fasting conditions in patients with and without T2D. The investigators will also assess how glucagon, a hormone that raises blood glucose levels, impacts the conversion of glycerol and lactate to glucose. Enrolled participants will undergo three separate isotope tracer infusions with serial blood collections for liquid chromatography-mass spectrometry analysis. This research could identify new therapeutic drug targets that can lower blood glucose levels more directly and effectively.

DETAILED DESCRIPTION:
Objectives:

1. Compare glycerol and lactate as carbon sources for GNG in humans with and without T2D.
2. Compare the contribution of glycerol and lactate to GNG during a hyperglucagonemic state.

Hypothesis:

1. Glycerol contributes to glucose and lactate production, while lactate is not a net carbon contributor to glucose or glycerol production.
2. Glycerol, not lactate, potentiates the observed increases in GNG seen in T2D.
3. Glucagon promotes greater glycerol incorporation into glucose as compared to lactate incorporation into glucose.

Study Design:

The investigators will recruit three different adult metabolic cohorts (16 per cohort): 1) Lean, defined as body mass index (BMI) <25.0 kg/m2, and no T2D; 2) Obese (BMI ≥ 30.0 kg/m2) and no T2D; and 3) Obese (BMI ≥ 30.0 kg/m2) and with T2D. All subjects will be between the ages of 18 and 65. All subjects will perform a self-monitored overnight fast at home and then come for three separate isotope tracer infusions (13C3-glycerol, 13C3-lactate, and 13C6-glucose) with serial blood draws. Each tracer infusion will last eight hours. During the final two hours of the infusion, subjects will receive intravenous glucagon, which increases the amount of glucose the liver produces. Collected blood samples will undergo liquid chromatography-mass spectrometry (LC-MS) analysis in our laboratory. Additionally, all subjects will receive a body composition analysis via dual-energy X-ray absorptiometry (DXA).

ELIGIBILITY:
Inclusion Criteria for All Subjects

1. Age 40-70 years.
2. The subject is otherwise in general good health, based on medical history and physical examination.

Inclusion Criteria for Metabolically Healthy Subjects without Obesity

1. No evidence of T2D or prediabetes as indicated by the American Diabetes Association (ADA), i.e., HbA1c < 5.7%, fasting glucose < 100 mg/dL, or use of glucose-lowering medications.
2. Body mass index (BMI) ≤ 24.9 kg/m2.

Inclusion Criteria for Metabolically Healthy Subjects with Obesity

1. No evidence of T2D or prediabetes as per ADA criteria.
2. 30.0 ≤ BMI ≤ 45.0 kg/m2.

Inclusion Criteria for T2D Subjects

1. Evidence of T2D as indicated by ADA criteria.
2. 6.5% ≤ HbA1c ≤ 8.0%.
3. 30.0 ≤ BMI ≤ 45.0 kg/m2.

Exclusion Criteria for All Subjects

1. Chronic medical conditions that may affect glucose metabolism, including active malignancy, tobacco use, HIV infection, kidney failure, liver dysfunction, alcoholism, pancreatitis, active viral/bacterial infection, current pregnancy/lactation, anemia, severe cardiac or respiratory failure, and uncontrolled hyperlipidemia (total cholesterol ≥ 260 mg/dL or triglycerides ≥400 mg/dL).
2. Current medical therapy that affects glucose metabolism such as glucocorticoid, antipsychotic, or oral contraceptive pills.
3. Type 1 diabetes mellitus diagnosis and/or history of diabetic ketoacidosis.
4. Use of weekly glucagon-like peptide-1 (GLP-1) receptor agonist therapy.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Carbon Contribution to Glucose Production | 8 hours
  Net carbon flux from glycerol and lactate to glucose will be measured using LC-MS of plasma glucose via 13C-enrichment after infusion of various metabolic tracers

CONTACTS AND LOCATIONS:
Overall Officials: Ankit Shah, MD, Principal Investigator — Rutgers Robert Wood Johnson Medical School

IPD SHARING:
Plan to Share IPD: No
Final data to be shared with study sponsor